CLINICAL TRIAL: NCT04080765
Title: Prospective Validation Study of a Antiretroviral Therapy (ARV) Decision Support Tool
Brief Title: Antiretroviral Therapy Selection: Comparing HIV Clinical Guidelines With HIV-ASSIST, an Online Decision-support Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00174416
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Hiv
Keywords: decision analysis; HIV; education
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-ASSIST + DHHS arm (Experimental): Decision-making support for ARV selection through DHHS guidelines in conjunction with HIV-ASSIST
  Interventions: Behavioral: HIV-ASSIST; Behavioral: DHHS guidelines
- DHHS-alone arm (Active Comparator): Decision-making support for ARV selection through DHHS guidelines alone
  Interventions: Behavioral: DHHS guidelines

INTERVENTIONS:
Behavioral: HIV-ASSIST — HIV-ASSIST is an online interactive patient-based tool that allows for individualized HIV treatment recommendations through the synthesis of patient-specific factors with existing guidelines and evidence.
  Arms: HIV-ASSIST + DHHS arm
Behavioral: DHHS guidelines — This is the Department of Health and Human Services HIV/AIDS Treatment Guidelines.

SUMMARY:
HIV-ASSIST is an online decision support tool created by Johns Hopkins faculty that utilizes standard patient variables, and provides treatment recommendations and tailored educational content to assist providers learn HIV treatment principles and support decision-making.

The research goal is to determine the difference in percentage of appropriate antiretroviral therapy (ART) selection (based upon a reference standard of HIV experts and guidelines) for a set of hypothetical patient scenarios, comparing a group of trainees with access to current national DHHS guidelines (control), and a group using HIV-ASSIST (intervention) in addition to guidelines.

The investigators proposed a randomized study design, in which an electronic survey/questionnaire with 10 HIV case vignettes are presented to study participants. Medical and nursing students and internal medicine residents will be eligible to participate.

Participants providing informed consent will be randomized to receiving access to either online Department of Health and Human Services (DHHS) HIV guidelines, or the HIV-ASSIST online tool to support participants' decision making. Participants will be asked to indicate participants' ART regimen of choice for each case scenario. The proportion of appropriate ART selections will be evaluated comparing the intervention and control arms. The investigators will additionally report the time required for trainees to complete ART selections for the presented clinical vignettes.

ELIGIBILITY:
Inclusion Criteria:

* Students in the Johns Hopkins Schools of Medicine or Nursing, and/or internal medicine residents

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-07-14 (Actual)

PRIMARY OUTCOMES:
Proportion of appropriate ARV selections | Up to one hour
  Median score (out of 100%) on survey of 10 standardized case scenarios, as scored in comparison to a reference panel of HIV experts.

SECONDARY OUTCOMES:
Time to ARV selection | Up to one hour
  Time in minutes to ARV selection for standardized case scenarios between trainees using HIV-ASSIST and those using the DHHS guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Maunank Shah, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez JA, Maddali MV, Nematollahi S, Li JZ, Shah M. New Strategies in Clinical Guideline Delivery: Randomized Trial of Online, Interactive Decision Support Versus Guidelines for Human Immunodeficiency Virus Treatment Selection by Trainees. Clin Infect Dis. 2021 May 4;72(9):1608-1614. doi: 10.1093/cid/ciaa299. PMID 32211758

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04080765/Prot_SAP_000.pdf